CLINICAL TRIAL: NCT03405610
Title: A Randomized Controlled Trial Testing a Skills-Based Program Called "A Toolkit for Optimal Recovery" Delivered Via Secure Live Video Compared to Standard Medical Care in Patients With Acute Musculoskeletal Injuries
Brief Title: A Skills-Based Program Delivered Via Secure Live Video to Patients With Acute Musculoskeletal Trauma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Ana-Maria Vranceanu, PhD, Clinical Psychologist, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2014P001194
Record Dates: First submitted 2017-12-03; First posted 2018-01-23 (Actual); Last update posted 2018-08-17 (Actual); Status verified 2018-08

CONDITIONS: Musculoskeletal Injury; Fracture
Keywords: Psychiatry; Psychology; Psychosocial; Mind-Body
MeSH Terms: conditions — Fractures, Bone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Toolkit for Optimal Recovery after Injury (Experimental): The Toolkit for Optimal Recovery after Injury (ToR) is a mind body skills based program delivered individually via secure live video. The format is a 4-week program with weekly meetings and a focus on teaching skills to optimize recovery and prevent chronic pain and disability.
  Interventions: Behavioral: The Toolkit for Optimal Recovery after Injury
- Usual Care (No Intervention): The Usual Care (UC) group will continue with their current medical care.

INTERVENTIONS:
Behavioral: The Toolkit for Optimal Recovery after Injury — The Toolkit for Optimal Recovery after Injury (ToR) is a skills based mind body program that was designed to prevent the development of chronic pain and disability following an acute musculoskeletal injury (e.g., fracture). The program has 4 sessions and it is delivered via live video. Patients learn myth about recovery after injury, false and real pain alarms, the fear avoidance model and how to prevent the disability spiral, mindfulness based exercises and activity pacing.
  Other Names: ToR
  Arms: Toolkit for Optimal Recovery after Injury

SUMMARY:
The aims of this study are to test a manualized mind body skills-building program aimed at preventing the development of chronic pain and disability following acute musculoskeletal injury in at-risk patients.

DETAILED DESCRIPTION:
This is a pilot randomized feasibility trial of the mind body program Toolkit for Optimal Recovery versus usual medical care. The Toolkit is delivered via secure live video to patients at risk for chronic pain, at 1-2 months after injury. The primary aim of this study is to determine the feasibility and acceptability of the program, randomization, procedures and outcome measures. Secondarily, we report means and standard deviation and explore change in quantitative outcomes in the Toolkit compared to usual care.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of musculoskeletal injury in the past 1-2 months
* 18 years of age or older
* English fluency and literacy
* PCS OR, PASS score above median split

Exclusion Criteria:

* Major medical comorbidity expected to worsen in the next 6 months
* Comorbid chronic pain condition
* Antidepressant medication change in the past 6 months
* Secondary gains such as litigations or workers compensation procedures
* Diagnosis of psychosis, bipolar disorder or active substance dependence (by self report)
* Unwilling or unable to use videoconferencing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2015-07-01 (Actual); Primary Completion 2018-08-01 (Actual); Study Completion 2018-08-01 (Actual)

PRIMARY OUTCOMES:
Feasibility of recruitment | 0 Weeks
  We will report number of patients approached, number who agreed to participate/were screened, number of patients randomized
Satisfaction with ToR | 4 weeks; 3 months
  3 questions assessing satisfaction with the physical recovery, with the care delivered, and with the clinician.
Acceptability | 4 weeks; 3 months
  We will report number of patients who finished ToR and UC and completed post-test from those who started the study (were randomized); We will also report number of participants who provided 3 months follow up
Feasibility of outcome measures | 0 weeks; 4 weeks; 3 months
  We will report number of missing items and calculate reliability of outcome measures
Adherence to ToR | 4 weeks.
  We will report number of participants who completed at least 3 out of 4 ToR sessions
Adherence to homework | 4 weeks
  determined by number of homework logs returned
Therapist adherence survey | 4 weeks
  Items assessing whether the therapist taught each of the skills included in each of the 4 sessions

SECONDARY OUTCOMES:
Pain Catastrophizing | 0 Weeks, 4 Weeks, 3 Months
  Pain Catastrophizing Scale (PCS); items are summed to generate a total score; scores range from 0 to 52; higher scores indicate greater pain catastrophizing
Pain Anxiety | 0 Weeks, 4 Weeks, 3 Months
  Pain Anxiety Symptom Scale (PASS); items are summed to generate a total score; scores range from 0-100; higher sores indicate greater pain anxiety
Depression | 0 Weeks, 4 Weeks, 3 Months
  Center for Epidemiologic Studies Depression Scale (CESD); items are summed to generate a total score; scores range from 0 to 60; higher scores indicate greater depressive symptomatology
Post Traumatic Stress Disorder | 0 Weeks, 4 Weeks, 3 Months
  Post Traumatic Stress Disorder Checklist (PCL); items are summed to generate a total score; scores range from 17 to 85; higher scores indicate greater post traumatic stress
Pain intensity | 0 Weeks, 4 Weeks, 3 Months
  Numerical rating scale assessing pain form 0 to 10
Physical Function | 0 Weeks, 4 Weeks, 3 Months
  Short Musculoskeletal Function Assessment (SMFA); two scores are generated by summing items 1-34 for Function Index and 35-46 for Bothersome Index;

CONTACTS AND LOCATIONS:
Overall Officials: Ana-Maria Vranceanu, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Vranceanu AM, Jacobs C, Lin A, Greenberg J, Funes CJ, Harris MB, Heng MM, Macklin EA, Ring D. Results of a feasibility randomized controlled trial (RCT) of the Toolkit for Optimal Recovery (TOR): a live video program to prevent chronic pain in at-risk adults with orthopedic injuries. Pilot Feasibility Stud. 2019 Feb 20;5:30. doi: 10.1186/s40814-019-0416-7. eCollection 2019. PMID 30820341